CLINICAL TRIAL: NCT04742712
Title: A Feasibility Study Using the CoronaCheck Device to Identify Incident Cases of SARS CoV-2 - FIND SARS CoV-2 Covid-19
Brief Title: A Feasibility Study Using the CoronaCheck Device to Identify Incident Cases of SARS CoV-2 Covid-19
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2020/57
Record Dates: First submitted 2020-10-28; First posted 2021-02-08 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: SARS-CoV Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RT-PCR swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CoronaCheck Device — All participants breath normally into the device for up to 6 minutes

SUMMARY:
Point of care testing is urgently required to enable the immediate detection of SARS-CoV-2 infection to allow effective transmission prevention precautions to succeed.

DETAILED DESCRIPTION:
The Coronacheck device is a hand-held, portable, point-of-care device which will allow the safe collection of EBC. It provides an automated platform for the detection of SARS-CoV-2 using an existing sensor repurposed with immobilised recombinant ACE-2 to bind the virus. This produces a measurable signal indicating whether SARS-CoV-2 is present or not.

EBC is collected by the CoronaCheck device during tidal breathing, making this investigation non-invasive, repeatable and easy to perform. Previous studies using Inflammacheck™ in people with respiratory conditions have shown it is well tolerated, even in people with severe lung disease. The full test cycle including sample collection and test assay typically occurs in less than 5 minutes.

Given the risk of infection, this CoronaCheck™ device has an integrated sensor and breath collection system combined in a fully enclosed, disposable unit to mitigate the risk of cross-infections between users and also reduces any exposure risk to healthcare staff. It is appreciated that disposable plastic has a negative environmental impact, however due to the highly contagious nature of SARS-CoV-2 it is felt unavoidable at present.

Using the CoronaCheck does not require laboratory equipment or expertise, and is a quick, easy-to-use point-of-care investigation which provides an immediate result. This could potentially be applied to screening for SARS-CoV-2 in a wide variety of environments for example: GP practices, drive-thru centres, colleges, universities, airports and sports arenas.

Any person undergoing a swab for a possible SARS CoV-2 infection is eligible for inclusion, participants will not be assigned an intervention.

The participants will breathe into the CoronaCheck device. This involves breathing for up to 6 minutes into a single use, fully sealed unit attached to the hand-held device. This disposable unit has a bacterial-viral filter attached to both the breathing inlet and the exhale outlet to eliminate any risk of contamination. The CoronaCheck device then provides a reading reflecting EBC ACE2 binding which will be documented on the eCRF. This result will not be recorded in the clinical notes as it is not intended to inform patient management decisions in this study.

ELIGIBILITY:
Inclusion Criteria:

o Any adult (≥ 16 years of age) who is:

* undergoing a swab for possible SARS-CoV-2 infection
* willing and able to give informed consent for participation in the study
* unlikely to suffer harm as a result of testing in the opinion of the investigator

Exclusion Criteria:

o Participants receiving:

* invasive ventilation, non-invasive ventilation or nasal high flow oxygen
* supplementary oxygen with symptomatic hypoxia or oxygen saturations ≤92% (≤88% in COPD) despite 4L oxygen via nasal cannulae
* unable to comprehend the study or provide informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A cross-sectional study including four groups at different stages of the diagnostic and screening process for potential SARS-CoV-2 infection, utilising RT-PCR from nasopharyngeal swab as the current gold standard:
  1. Participants with clinically suspected SARS-CoV-2 confirmed with a positive RT-PCR swab (inpatient or outpatient testing)
  2. Participants with clinically suspected SARS-CoV-2 but a negative RT-PCR swab (inpatient or outpatient testing)
  3. Asymptomatic participants with a low clinical suspicion of SARS-CoV-2 but a positive RT-PCR swab
  4. Asymptomatic participants with a low clinical suspicion of SARS-CoV-2 and a negative RT-PCR swab
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Presence of SARS-CoV-2 infection in those with high clinical suspicion and/or a positive RT-PCR swab. | through study completion, an average of 1 year
  Measured using the CoronaCheck device

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No